CLINICAL TRIAL: NCT05712395
Title: The Effects of a Novel, Non-ischemic and Pain-free Exercise Intervention in Peripheral Artery Disease
Acronym: NICE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Case Western Reserve University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16294; R01AG071778-01A1 (NIH)
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Claudication; Peripheral Artery Disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-Ischemic Exercise (NICE) exercise program (Experimental): Patients will perform supervised treadmill walking for 3 months. Patients randomized to the NICE program will walk intermittently at a slow speed of approximately 1.4 mph for only 2-3 minute bouts that do not elicit claudication pain.
  Interventions: Behavioral: Exercise
- Standard exercise program (Active Comparator): Patients will perform supervised treadmill walking for 3 months. Patients randomized to the Standard program will walk intermittently at a speed of approximately two mph to near maximal claudication pain.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Non-Ischemic Exercise (NICE), pain-free exercise program will be compared to the Standard painful exercise program.

SUMMARY:
This study is a 3-month, prospective, randomized controlled clinical trial designed to address the efficacy of the Non-Ischemic Exercise (NICE) program to improve exercise and vascular outcome measures in patients with peripheral artery disease (PAD).

DETAILED DESCRIPTION:
Specific Aims. The investigator proposes to test our central hypothesis that the NICE intervention performed without inducing leg ischemia and its' damaging sequela will be a superior exercise paradigm to increase peak walking time and HRQoL more than the Standard ischemic and painful exercise paradigm via greater improvement in microvascular mechanisms. This clinically relevant hypothesis will be tested through the following aims:

Aim 1 (Exercise Outcomes) To compare the changes in ambulation and HRQoL in PAD patients randomized to either the NICE slow walking program or to the Standard program of ischemic and painful exercise.

Aim 2a (Vascular Outcomes) To compare the changes in local microvascular function of the lower extremities, inflammation and oxidative stress in patients following the NICE program, and following the Standard ischemic and painful program.

Aim 2b (Exploratory Aim) To explore whether the changes in local microvascular function and systemic vascular biomarkers are associated with the changes in peak walking time following the NICE and Standard programs, and whether the association is stronger following the NICE program.

Methods. This is a 3-month, patient-oriented, translational, comparative effectiveness randomized controlled trial. One-hundred patients will be randomized into either the NICE program (N=50) or the Standard exercise program (N=50). All patients will perform supervised treadmill walking for 3 months. Patients randomized to the NICE program will walk intermittently at a slow speed of approximately 1.4 mph for only 2-3 minute bouts that do not elicit claudication pain. Patients randomized to the Standard program will walk intermittently at a speed of approximately two mph to near maximal claudication pain.

ELIGIBILITY:
Inclusion Criteria:

1. history of claudication assessed by the Walking Impairment Questionnaire,
2. ambulatory leg pain in either one or both legs consistent with intermittent claudication confirmed during a screening graded treadmill test using the Gardner-Skinner protocol,
3. an ABI <= 0.90 at rest or > 20% decrease in ankle systolic blood pressure in either one or both legs immediately following the treadmill exercise test.
4. age >= 60 years.

Exclusion Criteria:

1. absence of PAD (ABI > 0.90 at rest and ankle systolic blood pressure < 20% decrease after exercise,
2. inability to obtain an ABI measure due to non-compressible vessels (ABI > 1.40),
3. asymptomatic PAD (Fontaine Stage I) determined from the medical history and verified during the graded treadmill test,
4. rest pain due to PAD (Fontaine stage III)
5. tissue loss due to PAD (Fontaine stage IV)
6. use of medications indicated for the treatment of intermittent claudication (cilostazol and pentoxifylline) initiated within three months prior to investigation,
7. peripheral revascularization within one month prior to investigation, or peripheral revascularization performed during the study,
8. exercise tolerance limited by any disease process other than PAD,
9. active cancer,
10. kidney failure defined as stage 5 chronic kidney disease,
11. a calf skin fold measurement > 25 mm, because of potential interference with the light path of the NIRS probe from penetrating the subcutaneous tissue,
12. pulse arterial oxygen saturation of the index finger < 95% because of potential deleterious effect on calf muscle StO2 from poor pulmonary gas exchange, and
13. failure to complete the baseline run-in phase within three weeks.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2029-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Peak Walking Time | 3 months
  The change in peak walking time from the pre-test value to the post-test value (seconds)
Calf Muscle Oxygen Saturation | 3 months
  The change in calf muscle oxygen saturation value during exercise from the pre-test value to the post-test value (% saturation)

SECONDARY OUTCOMES:
6-Minute Walk Distance | 3 months
  The change in 6-minute walk distance from the pre-test value to the post-test value (meters)
plasma C-Reactive Protein | 3 months
  The change in plasma C-reactive protein from the pre-test value to the post-test value (mg/L)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W. Gardner, Ph.D, Principal Investigator — Professor, Department of Medicine, Cardiology
Locations (1):
- O'Donoghue Research Building, University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gardner AW, Parker DE, Montgomery PS, Scott KJ, Blevins SM. Efficacy of quantified home-based exercise and supervised exercise in patients with intermittent claudication: a randomized controlled trial. Circulation. 2011 Feb 8;123(5):491-8. doi: 10.1161/CIRCULATIONAHA.110.963066. Epub 2011 Jan 24. PMID 21262997
- [Result] Gardner AW, Parker DE, Montgomery PS, Blevins SM. Step-monitored home exercise improves ambulation, vascular function, and inflammation in symptomatic patients with peripheral artery disease: a randomized controlled trial. J Am Heart Assoc. 2014 Sep 18;3(5):e001107. doi: 10.1161/JAHA.114.001107. PMID 25237048